CLINICAL TRIAL: NCT01208740
Title: Effects of Metformin on the Ovarian Response to Gonadotropins for in Vitro Fertilization Treatment in Patients With Polycystic Ovary Syndrome and Predictors of Poor Ovarian Response
Brief Title: Metformin in Patients With PCOS and Predictors of Poor Ovarian Response Ongoing In-vitro Fertilization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Concerns about safety at the first interim analysis
Sponsor: University Magna Graecia (Other)
Responsible Party: Department of Obstetrics and Gynecology, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02/2010
Record Dates: First submitted 2010-05-24; First posted 2010-09-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Infertility; PCOS; Prognosis for Poor Response
Keywords: Gonadotropins; infertility; IVF; metformin; PCOS; poor prognosis; poor responder
MeSH Terms: conditions — Infertility | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin pre-treatment and co-administration
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo pre-treatment and co-administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500 mg three times daily
  Arms: Metformin
Drug: Placebo — 1 pill three times daily
  Arms: Placebo

SUMMARY:
Metformin should be administered with caution and could be potentially dangerous in infertile patients with PCOS who show a poor ovarian response and are undergoing gonadotropin-based ovarian stimulation. However, data that address this point are totally lacking.

On the basis of these considerations, the aim of the current clinical trial was to test the hypothesis that metformin reduces the ovarian response in infertile patients with PCOS who have a potentially poor ovarian response and who undergo gonadotropin stimulation for IVF cycles.

DETAILED DESCRIPTION:
Primary infertile patients with PCOS older than 35 years and/or with a basal follicle-stimulating hormone (FSH) level higher than 10 IU/L who were scheduled for IVF cycles were enrolled in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Prognosis for poor response
* Infertility

Exclusion Criteria:

* Male factor infertility
* Tubal infertility

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Rate of cancellation due to low ovarian response | one month
  Number of cancelled cycles/total cycles

SECONDARY OUTCOMES:
Stimulation length | one month
Gonadotropins dose | one month
Ovulation rate | one month
pregnancy rate | one month
Live-birth rate | nine months
Adverse effects | one month

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, MD, Study Chair — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- Pugliese" Hospital, Catanzaro, Italy, Italy

REFERENCES:
- [Derived] Palomba S, Falbo A, Di Cello A, Cappiello F, Tolino A, Zullo F. Does metformin affect the ovarian response to gonadotropins for in vitro fertilization treatment in patients with polycystic ovary syndrome and reduced ovarian reserve? A randomized controlled trial. Fertil Steril. 2011 Nov;96(5):1128-33. doi: 10.1016/j.fertnstert.2011.08.020. Epub 2011 Sep 13. PMID 21917254